CLINICAL TRIAL: NCT06778044
Title: Evaluation of an Online Self-Help Program for CSAM
Brief Title: ReDirection / Self-Guided ICBT to Reduce the Risk of Child Sexual Abuse Material (CSAM) Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); Protect Children Organisation, Finland (Unknown)
Responsible Party: Principal Investigator, Carissa Augustyn, Principal Investigator, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0246; OFIL-20-257 (Other Grant/Funding Number: Oak Foundation)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Pedophilia
Keywords: Child Sexual Abuse Material; Paraphilic Disorders; Waitlist; Child sexual abuse; Cognitive behavioural therapy; Self-help intervention; Internet based intervention; Prevention; Pedophilic disorder
MeSH Terms: conditions — Pedophilia; Paraphilic Disorders | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: A three-arm randomized controlled trial where two treatment arms (ReDirection 1.0 and ReDirection 2.0) are compared to a waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ReDirection 1.0 (Experimental)
  Interventions: Other: ReDirection 1.0
- ReDirection 2.0 (Experimental)
  Interventions: Other: ReDirection 2.0
- Waitlist (Active Comparator)
  Interventions: Other: Waitlist

INTERVENTIONS:
Other: ReDirection 1.0 — A free, anonymous, online, self-guided cognitive behavioral therapy (CBT) intervention. Consists of 6 modules.
  Arms: ReDirection 1.0
Other: ReDirection 2.0 — A free, anonymous, online, self-guided, cognitive behavioural therapy (CBT) intervention. Consists of 5 modules and the option for asynchronous messaging with a ReDirection specialist.
  Arms: ReDirection 2.0
Other: Waitlist — Participants in the waitlist control will wait six weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing sexual urges and behaviour.
  Arms: Waitlist

SUMMARY:
The creation and distribution of child sexual abuse material (CSAM) is a large-scale global problem. CSAM is sometimes referred to as child pornography. It includes images, videos, live-streaming, and any other material that depicts sexual acts with a child or adolescent (i.e., a person under the age of 18). It also includes material that shows a child or adolescent in a sexually suggestive or explicit manner partially clothed, or nude, and can include material that does or does not illustrate sexual activity.

CSAM use is a problem that continues to drastically increase in size despite the numerous political, police, and technological initiatives that have been put forth as solutions. Previous research also suggests that many active CSAM users desire help to stop their use, but have experienced difficulties finding support that is anonymous. Thus, there is a great need for anonymous intervention programs that assist active and at-risk CSAM users in developing skills to manage their thoughts, feelings, and behaviours related to CSAM.

ReDirection is a free, anonymous, online, self-guided, cognitive behavioural therapy (CBT)-based program for individuals concerned about their use or risk to use CSAM. The treatment program is based on many years of clinical experience working with patients who have committed sexual offences, and the results of several previous research projects.

This study will implement a scientifically rigorous design (a three-armed randomized waitlist-controlled trial) to evaluate two versions of this intervention (ReDirection 1.0 and ReDirection 2.0). The primary difference between the two versions of ReDirection is the length of the program and whether it includes the option for asynchronous messaging with a ReDirection specialist. The study design compares ReDirection 1.0 and ReDirection 2.0 with a waitlist control group. Participants in the waitlist control will wait six weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing about sexual urges and behaviours.

Participants will be recruited directly from the ReDirection website, where they will be directed to a secure platform designed specifically for clinical trials of internet-mediated CBT. This platform is called Iterapi. Potential participants learn about the ReDirection program through advertisements on both the "Clearnet" and "Darknet." All trial activities, including participant registration, random assignment, intervention, and evaluation will be conducted via Iterapi.

Treatment includes five-to-six modules over five-to-six weeks and the content includes CBT-based psychoeducation and exercises that aim to help participants gain greater understanding of, and skills to manage risky sexual thoughts, feelings, and behaviours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to read and understand English or Spanish
* Have used or experienced urges to use CSAM within the last six months

Exclusion Criteria:

* Younger than 18 years of age
* Unable to read and understand English or Spanish
* Have not used or experienced urges to use CSAM within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Do ReDirection 1.0 and ReDirection 2.0 reduce participants' urges to use CSAM? | Up to 8 weeks
  Urges to use CSAM is measured using a modified version of the SSAS (Sexual Symptom Assessment Scale), which is a self-rated measure originally developed to assess general sexual compulsive behaviour. This measure was adapted to include language specific to CSAM use, and response options were altered to permit more precise measurement.
  There's no scoring system at the moment. It's all item-by-item. But for all items, higher values indicated a greater frequency, intensity, and/or duration of urges.

SECONDARY OUTCOMES:
Do ReDirection 1.0 and ReDirection 2.0 reduce participants' proclivity to offend? | Up to 8 weeks
  Proclivity to offend is defined as likelihood to engage in offending behaviour if no one were to ever find out and the individual could not be punished. This is assessed using two separate items created for this study: one for likelihood of CSAM use and one for likelihood of sexual contact with a person 15 years of age or younger. These are each measured as a likelihood from 0 [minimum] to 100 [maximum]. A 0 indicates 'no chance' whereas 100 indicates 'guaranteed'

CONTACTS AND LOCATIONS:
Overall Officials: Carissa Augustyn, PhD, Principal Investigator — The Royal Ottawa Mental Health Centre
Locations (2):
- University of Ottawa Integrated Mental Health Research at The Royal, Ottawa, Canada
- Protect Children NGO, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in each respective article (text, tables, figures and appendices). Data will be shared with an approved data access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following each article publication.
Access Criteria: Investigators who provide a methodologically sound proposal, and whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  Proposals should be directed to carissa.augustyn@theroyal.ca. To gain access to the data , data requesters will need to sign a data access agreement. Data will be made available digitally via a secure data transfer.